CLINICAL TRIAL: NCT04586868
Title: VR-assisted Cognitive Behaviour Therapy for Adolescents With Psychosis
Brief Title: VR-assisted CBT for Adolescents With Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95428
Record Dates: First submitted 2020-09-16; First posted 2020-10-14 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-03

CONDITIONS: Psychotic Disorders
Keywords: Psychosis; Adolescents; Virtual Reality treatment; Cognitive Behavioural Therapy; Early onset psychosis; VR-assisted therapy
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A psychotic disorder (Experimental): Patients, age 13-18 years old, diagnosed with a psychotic disorder (WHO ICD-10 )
  Interventions: Behavioral: An intervention development study; Behavioral: A randomized feasibility study; Behavioral: A single-case study

INTERVENTIONS:
Behavioral: An intervention development study — Assessing the acceptability for a virtual reality intervention among adolescents with psychosis
Behavioral: A randomized feasibility study — Feasibility of virtual reality environment for adolescents with psychosis
Behavioral: A single-case study — The clinical efficacy of a novel VR-assisted CBT interventions for adolescents with psychosis

SUMMARY:
Psychotic disorders typically emerge during late adolescence or early adulthood. Patients, who are diagnosed with a psychotic disorder before turning 18 years, are defined as early onset psychosis patients (EOP). Relative to adult patients, these patients show a worse long-term prognoses. Social impairment present a major barrier towards recovery, and thus and important issue to address in treatment. Cognitive behavioral therapy (CBT) is the recommended psychological treatment for psychotic disorders. As part of the therapy, the patient does an exposure-based training in a social environment. This type of training has several limitations for patients with psychosis. The last decade there has been a growing interest in using virtual reality (VR) to understand and treat various psychological disorders. There is a lack of research on VR-interventions for EOP patients. This study will assess the acceptability, tolerability, feasibility and clinical efficacy of a novel VR-assisted CBT interventions for adolescents with psychosis.

DETAILED DESCRIPTION:
This study adhere to the model for research made by the international Virtual Reality Clinical Outcomes Research Experts groups (VR-CORE). The study consist of three sub-studies. First a qualitative study assessing the acceptability for VR among adolescence with psychosis. Secondly, a randomized study of the feasibility of virtual reality environment for adolescents with psychosis. Third, assessing the clinical efficacy of a novel VR-assisted CBT interventions for adolescents with psychosis, through a non-randomized single-case study.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from a psychotic disorder (ICD-10 WHO)
* In stable clinical condition (i.e. not hospitalized)
* Being able to speak Norwegian or a Scandinavian language, or English
* Able to provide informed consent.

Exclusion Criteria:

* Primary neurological or endocrinological disorder
* Started a "transfer-process" to Department of Adult Psychiatry.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability for a virtual reality intervention | 5 months
  Semi-structured interview
Social self-efficacy | 1 week before, and 10 minutes after treatment.
  Adolescent self-efficacy scale (S-EFF)
Social interaction and social phobia | 1 week before, and 10 minutes after treatment.
  Short Form Social Interaction Anxiety Scale/Social Phobia Scale (SIAS-6/SPS-6)
Social paranoia | 1 week before and 1 week after treatment.
  State Social Paranoia Scale (SSPS)

SECONDARY OUTCOMES:
Self-esteem | 1 week before, and 10 minutes after treatment.
  Rosenberg Self-Esteem scale (RSES)
Psychotic symptoms | 1 week before and 1 week after treatment.
  Brief Psychiatric Rating Scale (BPRS)
The experience of presence | 10 minutes after treatment
  Gatineau Presence Questionnaire (GPQ)
Unwanted side effect | 10 minutes before and 10 minutes after treatment
  Virtual Reality Sickness Questionnaire (VRSQ)

OTHER OUTCOMES:
Level of functioning | 1 week after treatment.
  Children's Global Assessment Scale (C-GAS)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Elgen, phd, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland university hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holgersen G, Nordgreen T, Ten Velden Hegelstad W, Bircow Elgen I. Views of young people with psychosis on using virtual reality assisted therapy. A qualitative study. Early Interv Psychiatry. 2023 Apr;17(4):361-367. doi: 10.1111/eip.13331. Epub 2022 Jun 16. PMID 35708166